CLINICAL TRIAL: NCT00479401
Title: A Double-blind, Double-dummy, Placebo-controlled, Randomized, Three Parallel Groups Study Comparing the Efficacy, Safety and Tolerability of Pramipexole ER Versus Placebo and Versus Pramipexole IR Administered Orally Over a 26-week Maintenance Phase in Patients With Early Parkinsons Disease (PD).
Brief Title: Efficacy, Safety, Tolerability of Pramipexol ER Versus Pramipexol IR Versus Placebo in Early PD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 248.524; Eudract No 2007-000073-39
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Results first posted 2010-04-15 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-06

CONDITIONS: Early Parkinson Disease (Early PD)
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Pramipexole Extended Release (PPX ER) (Experimental)
  Interventions: Drug: Pramipexol Extended Release
- Pramipexole Immediate Release (PPX IR) (Experimental)
  Interventions: Drug: Pramipexol Immediate Release
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pramipexol Extended Release
  Arms: Pramipexole Extended Release (PPX ER)
Drug: Pramipexol Immediate Release
  Arms: Pramipexole Immediate Release (PPX IR)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objectives of this trial conducted in early Parkinson's Disease (PD) patients are to determine the efficacy (as measured by the change from baseline to the end of the maintenance phase in the total score for the Unified Parkinson's Disease Rating Scale (UPDRS) Parts II and III combined), safety, and tolerability of Pramipexole Extended Release (ER) (in daily doses from 0.375mg to 4.5mg q.d.) in comparison to placebo, and to test for non-inferiority between the two formulations (ER and IR) of pramipexole.

In addition, the efficacy of Pramipexole Immediate Release (IR) will be compared to placebo, for assay sensitivity

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient with idiopathic Parkinsons disease (PD) confirmed by at least two of the following signs: resting tremor, bradykinesia, rigidity.
2. Parkinsons disease diagnosed within 5 years.
3. Patients 30 years of age or older at the time of diagnosis.
4. Modified Hoehn and Yahr stage of 1 to 3.
5. Patients requiring additional therapy/ introduction of therapy (for de novo patients) to treat their parkinsonian symptoms at the time of enrollment (screening visit, V1) according to the investigators judgement.

Exclusion Criteria:

1. Atypical parkinsonian syndromes due to drugs (e.g., metoclopramide, flunarizine), metabolic disorders (e.g., Wilson's disease), encephalitis or degenerative diseases (e.g., progressive supranuclear palsy).
2. Dementia, as defined by a Mini-Mental State Exam score < 24 at screening visit
3. Any psychiatric disorder according to Diagnostic and Statistical Manual of Mental Disorders 4th (DSM-IV)
4. History of psychosis
5. Clinically significant electrocardiogram (ECG) abnormalities at screening visit
6. Clinically significant hypotension
7. Malignant melanoma or history of previously treated malignant melanoma
8. Any other clinically significant disease, whether treated or not, that could put the patient at risk or could prevent compliance or completion of the study
9. Pregnancy
10. Sexually active female of childbearing potential not using a medically approved method of birth control
11. Serum levels of Aspartate Aminotransferase (AST) , Alanine Aminotransferase (ALT), alkaline phosphatases or bilirubin > 2 Upper Limit of Normal (ULN)
12. Patients with a creatinine clearance < 50 mL/min
13. Any dopamine agonist (including pramipexole) within 4 weeks prior to baseline visit, or L-Dopa within 8 weeks prior to baseline visit.
14. Total cumulative duration of prior exposure to Levodopa of more than 3 months.
15. Any medication (including intra-muscular formulations) with central dopaminergic antagonist activity within 4 weeks prior to the baseline visit
16. Any of the following drugs within 4 weeks prior to the baseline visit: methylphenidate, cinnarizine, amphetamines.
17. Flunarizine within 3 months prior to baseline visit
18. Known hypersensitivity to Pramipexole or its excipients
19. Drug abuse (including alcohol), according to Investigators judgement, within 2 years prior to screening.
20. Participation in other investigational drug studies or use of other investigational drugs within one month or five times the half-life of the investigational drug

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 539 (Actual)
Dates: Start 2007-05; Primary Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (95):
- United States (16):
  - 248.524.01018 Boehringer Ingelheim Investigational Site, Gilbert, Arizona
  - 248.524.01004 Boehringer Ingelheim Investigational Site, Sun City, Arizona
  - 248.524.01016 Boehringer Ingelheim Investigational Site, La Jolla, California
  - 248.524.01013 Boehringer Ingelheim Investigational Site, Oxnard, California
  - 248.524.01008 Boehringer Ingelheim Investigational Site, Danbury, Connecticut
  - 248.524.01010 Boehringer Ingelheim Investigational Site, Boca Raton, Florida
  - 248.524.01014 Boehringer Ingelheim Investigational Site, Augusta, Georgia
  - 248.524.01012 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 248.524.01001 Boehringer Ingelheim Investigational Site, Kansas City, Kansas
  - 248.524.01007 Boehringer Ingelheim Investigational Site, Elkridge, Maryland
  - 248.524.01015 Boehringer Ingelheim Investigational Site, Southfield, Michigan
  - 248.524.01017 Boehringer Ingelheim Investigational Site, Hattiesburg, Mississippi
  - 248.524.01005 Boehringer Ingelheim Investigational Site, Commack, New York
  - 248.524.01002 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 248.524.01003 Boehringer Ingelheim Investigational Site, Midvale, Utah
  - 248.524.01009 Boehringer Ingelheim Investigational Site, Burlington, Vermont
- Argentina (8):
  - 248.524.54001 Boehringer Ingelheim Investigational Site, Capital Federal
  - 248.524.54002 Boehringer Ingelheim Investigational Site, Capital Federal
  - 248.524.54003 Boehringer Ingelheim Investigational Site, Capital Federal
  - 248.524.54007 Boehringer Ingelheim Investigational Site, Capital Federal
  - 248.524.54008 Instituto de Neurociencias de Buenos Aires, Capital Federal
  - 248.524.54009 Boehringer Ingelheim Investigational Site, Capital Federal
  - 248.524.54006 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 248.524.54004 Boehringer Ingelheim Investigational Site, Santa Fe
- Austria (2):
  - 248.524.43001 Boehringer Ingelheim Investigational Site, Innsbruck
  - 248.524.43004 Boehringer Ingelheim Investigational Site, Vienna
- Czechia (4):
  - 248.524.42004 Boehringer Ingelheim Investigational Site, Olomouc
  - 248.524.42003 Boehringer Ingelheim Investigational Site, Pardubice
  - 248.524.42001 Boehringer Ingelheim Investigational Site, Prague
  - 248.524.42002 Boehringer Ingelheim Investigational Site, Rychnov nad Kněžnou
- Finland (3):
  - 248.524.35803 Boehringer Ingelheim Investigational Site, Hyvinkää
  - 248.524.35801 Boehringer Ingelheim Investigational Site, Oulu
  - 248.524.35802 Boehringer Ingelheim Investigational Site, Tampere
- Germany (9):
  - 248.524.49002 Boehringer Ingelheim Investigational Site, Berlin
  - 248.524.49003 Boehringer Ingelheim Investigational Site, Bochum
  - 248.524.49011 Boehringer Ingelheim Investigational Site, Bochum
  - 248.524.49008 Boehringer Ingelheim Investigational Site, Bremerhaven
  - 248.524.49006 Boehringer Ingelheim Investigational Site, Dresden
  - 248.524.49007 Boehringer Ingelheim Investigational Site, Göttingen
  - 248.524.49001 Boehringer Ingelheim Investigational Site, Kassel
  - 248.524.49004 Boehringer Ingelheim Investigational Site, Leipzig
  - 248.524.49005 Boehringer Ingelheim Investigational Site, Marburg
- Hungary (8):
  - 248.524.36007 Boehringer Ingelheim Investigational Site, Eger
  - 248.524.36005 Boehringer Ingelheim Investigational Site, Győr
  - 248.524.36008 Boehringer Ingelheim Investigational Site, Miskolc
  - 248.524.36004 Boehringer Ingelheim Investigational Site, Sopron
  - 248.524.36001 Boehringer Ingelheim Investigational Site, Szeged
  - 248.524.36006 Boehringer Ingelheim Investigational Site, Szeged
  - 248.524.36003 Boehringer Ingelheim Investigational Site, Szombathely
  - 248.524.36002 Boehringer Ingelheim Investigational Site, Zalaegerszeg
- India (9):
  - 248.524.91002 Boehringer Ingelheim Investigational Site, Chennai
  - 248.524.91009 Boehringer Ingelheim Investigational Site, Hyderabad
  - 248.524.91010 Boehringer Ingelheim Investigational Site, Hyderabad
  - 248.524.91001 Boehringer Ingelheim Investigational Site, Karnataka
  - 248.524.91005 Boehringer Ingelheim Investigational Site, Maharashtra
  - 248.524.91007 Boehringer Ingelheim Investigational Site, Maharashtra
  - 248.524.91004 Boehringer Ingelheim Investigational Site, New Delhi
  - 248.524.91006 Boehringer Ingelheim Investigational Site, New Delhi
  - 248.524.91011 Boehringer Ingelheim Investigational Site, Pune
- Japan (15):
  - 248.524.81010 Boehringer Ingelheim Investigational Site, Aomori, Aomori
  - 248.524.81001 Boehringer Ingelheim Investigational Site, Bunkyo-ku, Tokyo
  - 248.524.81005 Boehringer Ingelheim Investigational Site, Fuchu, Tokyo
  - 248.524.81011 Boehringer Ingelheim Investigational Site, Fujisawa, Kanagawa
  - 248.524.81013 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 248.524.81015 Boehringer Ingelheim Investigational Site, Iwamizawa,Hokkaido
  - 248.524.81003 Boehringer Ingelheim Investigational Site, Kodaira, Tokyo
  - 248.524.81014 Boehringer Ingelheim Investigational Site, Kyoto, Kyoto
  - 248.524.81009 Boehringer Ingelheim Investigational Site, Morioka, Iwate
  - 248.524.81008 Boehringer Ingelheim Investigational Site, Okayama, Okayama
  - 248.524.81006 Boehringer Ingelheim Investigational Site, Ota-ku, Tokyo
  - 248.524.81004 Boehringer Ingelheim Investigational Site, Sagamihara, Kanagawa
  - 248.524.81007 Boehringer Ingelheim Investigational Site, Shimogyo-ku, Kyoto, Kyoto
  - 248.524.81012 Boehringer Ingelheim Investigational Site, Shiroishi, Miyagi
  - 248.524.81002 Boehringer Ingelheim Investigational Site, Takamatsu, Kagawa
- Malaysia (3):
  - 248.524.60001 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 248.524.60004 Boehringer Ingelheim Investigational Site, Kuala Terengganu
  - 248.524.60002 Boehringer Ingelheim Investigational Site, Pulau Pinang
- Russia (6):
  - 248.524.07001 Boehringer Ingelheim Investigational Site, Moscow
  - 248.524.07002 Boehringer Ingelheim Investigational Site, Moscow
  - 248.524.07003 Boehringer Ingelheim Investigational Site, Moscow
  - 248.524.07004 Boehringer Ingelheim Investigational Site, Moscow
  - 248.524.07005 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 248.524.07006 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Slovakia (2):
  - 248.524.42103 Boehringer Ingelheim Investigational Site, Dubnica nad Váhom
  - 248.524.42101 Boehringer Ingelheim Investigational Site, Trnava
- Taiwan (4):
  - 248.524.88603 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 248.524.88605 Boehringer Ingelheim Investigational Site, Taichung
  - 248.524.88601 Boehringer Ingelheim Investigational Site, Taipei
  - 248.524.88602 Boehringer Ingelheim Investigational Site, Taoyuan District
- Ukraine (6):
  - 248.524.38005 Boehringer Ingelheim Investigational Site, Kiev
  - 248.524.38001 Boehringer Ingelheim Investigational Site, Lviv
  - 248.524.38002 Boehringer Ingelheim Investigational Site, Uzhhorod
  - 248.524.38003 Boehringer Ingelheim Investigational Site, Vinnytzya
  - 248.524.38004 Boehringer Ingelheim Investigational Site, Zaporizhzhya
  - 248.524.38006 Boehringer Ingelheim Investigational Site, Zaporizhzhya

REFERENCES:
- See also: Related Info — http://trials.boehringer-ingelheim.com/content/dam/internet/opu/clinicaltrial/com_EN/results/248/248.524_Literature.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Pramipexole Extended Release (PPX ER): PPX ER tablets taken once in the morning
- Pramipexole Immediate Release (PPX IR): PPX IR tablets taken three times a day
- Placebo: Placebo to PPX ER once and to PPX IR three times a day
Period: Overall Study
Arm/Group | Pramipexole Extended Release (PPX ER) | Pramipexole Immediate Release (PPX IR) | Placebo
Started | 223 | 213 | 103
Completed | 174 | 176 | 91
Not Completed | 49 | 37 | 12
Not completed — Adverse Event | 24 | 20 | 4
Not completed — Lack of Efficacy | 2 | 2 | 4
Not completed — Protocol Violation | 2 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Withdrawal by Subject | 16 | 10 | 2
Not completed — Exclusion criteria, relocation | 4 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pramipexole Extended Release (PPX ER) | Pramipexole Immediate Release (PPX IR) | Placebo | Total
Number analyzed (Participants) | 223 | 213 | 103 | 539
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.8) | 61.7 (9.6) | 62.0 (9.6) | 61.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 92 | 52 | 240
  Male | 127 | 121 | 51 | 299

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Parts II+III Total Score
Description: Activities of daily living are scored from 0-52 in UPDRS II, result of motor examination scored 0-108 in UPDRS III. A decrease in the score means improvement.
Time Frame: baseline and after 33 weeks treatment
Population: Full Analysis Set, all randomized patients, received at least one dose of study drug and provided any post baseline efficacy assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pramipexole Extended Release (PPX ER) | Pramipexole Immediate Release (PPX IR) | Placebo
Number analyzed (Participants) | 213 | 207 | 103
units on a scale | -8.6 [-9.9 to -7.2] | -8.8 [-10.2 to -7.4] | -3.8 [-5.9 to -1.8]
Statistical Analysis 1: Comparison: Pramipexole Extended Release (PPX ER) vs Pramipexole Immediate Release (PPX IR); A non-inferiority hypothesis (H0: μER - μIR < -3 vs. H1: μER - μIR ≥ -3) comparing pramipexole ER to pramipexole IR was tested using a non-inferiority margin of -3 points; Test type: Non-Inferiority or Equivalence — A non-inferiority hypothesis comparing pramipexole ER to pramipexole IR was to be tested using a non-inferiority margin of -3 points. The primary efficacy endpoint in UPDRS part II+III was the change from baseline (week 0) to week 33 on the UPDRS Parts II+III score combined. The statistical model was analysis of covariance, controlling for baseline UPDRS Part II+III. Fixed terms in the model were treatment, country, and UPDRS Part II+III score at baseline; ANCOVA; Null hypothesis was tested using an analysis of covariance model with α = 0.05 in full analysis set with last observation carried forward; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-2.2 to 1.7] — PPX ER non-inferior to PPX IR, if the lower limit of the confidence interval for the difference is higher than the non-inferiority margin of -3

2. Secondary Outcome: Percentage of Responders on the Clinical Global Impressions of Improvement (CGI-I) Scale
Description: Clinicians evaluation in a rating scale of 7 steps, 1 meaning very much improved to 7 meaning very much worse. Responders are the patients with 'much improved' and 'very much improved' on the scale
Time Frame: after 18 weeks of treatment compared to baseline
Population: Full Analysis Set 1, all randomized patients, received at least one dose of study drug and provided any post baseline efficacy assessment and completed 18 weeks of treatment or discontinued prematurely at the interim cut off date Apr 2008
Measure: Number; unit: Percentage of Participants
Arm/Group | Pramipexole Extended Release (PPX ER) | Pramipexole Immediate Release (PPX IR) | Placebo
Number analyzed (Participants) | 100 | 100 | 50
Percentage of Participants | 37 | 48 | 18

3. Secondary Outcome: Percentage of Responders on the Patients Global Impressions of Improvement (PGI-I) Scale
Description: Patient rated evaluation of the PD symptoms on a rating scale of 7 steps, 1 meaning very much better to 7 meaning very much worse. Responders are the patients with 'much better' and 'very much better' on the score.
Time Frame: after 18 weeks of treatment compared to baseline
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Pramipexole Extended Release (PPX ER) | Pramipexole Immediate Release (PPX IR) | Placebo
Number analyzed (Participants) | 101 | 101 | 50
Percentage of Participants | 35.6 | 23.8 | 12

4. Secondary Outcome: UPDRS II+III Responder Rate (at Least 20% Improvement)
Description: Responders are defined as at least 20% decrease in the UPDRS II+III score. UPDRS II+III ranges 0-160 scores from best to worse.
Time Frame: after 33 weeks treatment
Population: as for outcome 1
Measure: Number; unit: percentage of responders
Arm/Group | Pramipexole Extended Release (PPX ER) | Pramipexole Immediate Release (PPX IR) | Placebo
Number analyzed (Participants) | 213 | 207 | 103
percentage of responders | 68.5 | 65.7 | 48.5

5. Secondary Outcome: UPDRS Part I Change From Baseline
Description: UPDRS I evaluates mentation behaviour and mood with a total score of 0-16. Decrease in the scores means improvement
Time Frame: baseline and after 33 weeks treatment
Population: Full Analysis Set with (LOCF), all randomized patients, received at least one dose of study drug and provided any post baseline efficacy assessment
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Pramipexole Extended Release (PPX ER) | Pramipexole Immediate Release (PPX IR) | Placebo
Number analyzed (Participants) | 213 | 207 | 103
units on a scale | 0.0 [-1.0 to 0.0] | 0.0 [-1.0 to 0.0] | 0.0 [-1.0 to 0.0]

6. Secondary Outcome: UPDRS Part II Total Score
Description: UPDRS II evaluates activities of daily living in a score 0-52. Decrease of the score means improvement
Time Frame: after 33 weeks treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pramipexole Extended Release (PPX ER) | Pramipexole Immediate Release (PPX IR) | Placebo
Number analyzed (Participants) | 213 | 207 | 103
units on a scale | -2.2 [-2.6 to -1.7] | -2.4 [-2.9 to -2.0] | -0.9 [-1.5 to -0.3]

7. Secondary Outcome: UPDRS Part III Total Score
Description: UPDRS III is the result of a motor examination with the scores 0-108. A decrease in the scores means improvement
Time Frame: after 33 weeks treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pramipexole Extended Release (PPX ER) | Pramipexole Immediate Release (PPX IR) | Placebo
Number analyzed (Participants) | 213 | 207 | 103
units on a scale | -6.4 [-7.4 to -5.4] | -6.4 [-7.4 to -5.4] | -2.8 [-4.2 to -1.4]

8. Secondary Outcome: Beck's Depression Inventory Version I A
Description: The Beck's Depression Inventory (BDI) is a 21-item self-rating scale that was originally designed as an instrument to assess the intensity of depressive symptoms (sadness, pessimism, sense of failure, dissatisfaction, guilt, expectation of punishment, dislike of self, self-accusation, suicidal ideation, episodes of crying, irritability, social withdrawal, indecisiveness, changes in body image, retardation, insomnia, fatigability, loss of appetite and weight, somatic preoccupation, low level of energy). Each item is scored from 0 (absent) to 3 (severe). The patients select the score which best describes their status in the last 7 days. Since its introduction in 1961, its use has been extended (also to PD patients) and today it is used also as a screening instrument as well as an outcome measure in depression treatment trials. The total score sums the 21 individual items yielding a score that can range from zero (minimal depression) to 63 (severe depression).
Time Frame: after 33 weeks treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pramipexole Extended Release (PPX ER) | Pramipexole Immediate Release (PPX IR) | Placebo
Number analyzed (Participants) | 208 | 206 | 102
units on a scale | -2.0 [-2.7 to -1.3] | -2.7 [-3.4 to -2.0] | -2.1 [-3.1 to -1.2]

9. Secondary Outcome: Likert Scale for Pain Related to PD
Description: Patient assessed 11 units on a scale from 'no pain' to 'unbearable pain'. Decrease of the score means improvement
Time Frame: after 33 weeks treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pramipexole Extended Release (PPX ER) | Pramipexole Immediate Release (PPX IR) | Placebo
Number analyzed (Participants) | 208 | 206 | 102
units on a scale | -0.2 [-0.4 to 0.1] | -0.1 [-0.4 to 0.1] | 0.2 [-0.2 to 0.5]

10. Secondary Outcome: Parkinson's Disease Sleep Scale (PDSS)
Description: PDSS is a self-rated instrument addressing 15 commonly reported symptoms associated with sleep disturbance on 15 visual analogue scales (VAS: 0 to 10 cm) each ranging from worst score ('awful or always' at the left extremity to the best score ('excellent or never' at the right extremity) An increase in the score means improvement. Worst possible score 0, best score 150)
Time Frame: after 33 weeks treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pramipexole Extended Release (PPX ER) | Pramipexole Immediate Release (PPX IR) | Placebo
Number analyzed (Participants) | 207 | 205 | 101
units on a scale | 2.3 [-0.4 to 5.0] | 5.6 [2.8 to 8.4] | 5.6 [1.8 to 9.4]

11. Secondary Outcome: Change From Baseline in Parkinson's Disease Quality of Life Questionnaire Total Score
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health which patients consider to be adversely affected by the disease. Higher scores are consistently associated with more severe symptoms of the disease such as tremor and stiffness, while lower scores indicate a better perceived health status. The 8 domains include:
  * mobility (e.g. fear of falling when walking): 10 items
  * activities of daily living (e.g. difficulty cutting food): 6 items
  * emotional well-being (e.g. feelings of isolation): 6 items
  * stigma (e.g. social embarrassment): 4 items
  * social support: 3 items
  * cognition: 4 items
  * communication: 3 items
  * bodily discomfort: 3 items.
  A total score is calculated by summing the responses to the 39 individual items and the total ranges from 0 (no problem at all) to 156 (maximum level of problem). A negative change in the total score indicates improvement.
Time Frame: after 33 weeks treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pramipexole Extended Release (PPX ER) | Pramipexole Immediate Release (PPX IR) | Placebo
Number analyzed (Participants) | 195 | 199 | 98
units on a scale | -4.1 [-6.1 to -2.0] | -6.5 [-8.6 to -4.5] | -2.1 [-4.9 to 0.8]

12. Secondary Outcome: Change From Baseline in European Quality of Life Visual Analog Scale
Description: European Quality of Life Visual Analog Scale (EQ-5D VAS) is a 20 centimeter vertical analog scale assessing the patient's general health status with scores ranging from 0 (worst imaginable health) to 100 (perfect health). A positive change in the scale indicates improvement in health status.
Time Frame: after 33 weeks treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pramipexole Extended Release (PPX ER) | Pramipexole Immediate Release (PPX IR) | Placebo
Number analyzed (Participants) | 195 | 199 | 98
units on a scale | 4.0 [1.4 to 7.6] | 6.6 [3.9 to 9.2] | 3.2 [-0.4 to 6.9]

13. Secondary Outcome: Patients Who Started to Use L-Dopa Rescue Medication
Description: L-dopa could be introduced as rescue medication based upon the clinical judgement of the investigator. descriptive on the Full Analysis Set (FAS) population
Time Frame: from trial start on to any time before final assessment of the patient, up to 33 weeks
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Pramipexole Extended Release (PPX ER) | Pramipexole Immediate Release (PPX IR) | Placebo
Number analyzed (Participants) | 213 | 207 | 103
patients | 15 | 9 | 22

14. Secondary Outcome: Number of Patients With Treatment Emergent Abnormal Behaviour as Indicated by the Modified Minnesota Impulsive Disorders Interview (mMIDI Questionnaire)
Description: mMIDI is a semi-structured clinical interview to assess pathological gambling (12 questions, positive screen if patient answers 'yes' to question 1 and to at least 5 of the rest of the questions), compulsive buying (9 questions from 1a to 4c, positive screen if the patient answers 'yes' to 1a, 2a, 3a, and 4a) and compulsive sexual behaviour (4 questions, positive screen if patient answers 'yes' to question 1,2,3, or 4).
Time Frame: from trial start on to any time before final assessment of the patient, up to 33 weeks
Population: Treated Set (TS), all randomized patients, who were dispensed study medication and documented to have taken at least 1 dose of study medication.
Measure: Number; unit: patients
Arm/Group | Pramipexole Extended Release (PPX ER) | Pramipexole Immediate Release (PPX IR) | Placebo
Number analyzed (Participants) | 223 | 213 | 103
patients | 4 | 3 | 1

15. Secondary Outcome: Possible Clinically Significant Abnormal Laboratory Parameters
Description: The significant abnormality of values was based on standard criteria defined in appendix 16.1.10, LISTING 4 Criteria for clinically significant abnormalities based on normalized laboratory values.
Time Frame: baseline and after 33 weeks of treatment
Population: Treated Set Labs (TSLabs), all patients in TS with a clinical laboratory measurements at baseline and at the last visit.
Measure: Number; unit: participants
Arm/Group | Pramipexole Extended Release (PPX ER) | Pramipexole Immediate Release (PPX IR) | Placebo
Number analyzed (Participants) | 199 | 202 | 99
participants
  Haematocrit - decrease | 4 (9.8) | 3 (10.1) | 1 (10.7)
  Haemoglobin - decrease | 11 | 6 | 1
  Red blood cell ct. - decrease | 1 | 0 | 0
  White blood cell ct. - decrease | 1 | 0 | 0
  Neut., poly (segs) - decrease | 2 | 0 | 0
  Eosinophils - increase | 6 | 3 | 3
  Neut., poly (segs), absol. - decrease | 1 | 0 | 0
  Sodium - decrease | 5 | 5 | 0
  Potassium - increase | 3 | 1 | 0
  Chloride - decrease | 2 | 0 | 0
  Alkaline phosphatase - increase | 0 | 1 | 0
  GGT - increase | 3 | 1 | 0
  Glucose - decrease | 3 | 0 | 0
  Glucose - increase | 1 | 1 | 0
  Cholesterol, total - increase | 0 | 0 | 1
  Creatinine - increase | 0 | 0 | 1
  Triglyceride - increase | 9 | 3 | 5
  Uric acid - increase | 3 | 1 | 2

16. Secondary Outcome: Clinical Relevant Abnormal Findings in Vital Signs and Physical Examination as Reported in Adverse Events
Time Frame: baseline and after 33 weeks of treatment
Population: Treated set (TS)
Measure: Number; unit: participants
Arm/Group | Pramipexole Extended Release (PPX ER) | Pramipexole Immediate Release (PPX IR) | Placebo
Number analyzed (Participants) | 223 | 213 | 103
participants
  Hypertension | 6 | 7 | 5
  Orthostatic hypotension | 7 | 1 | 1
  Hypotension | 0 | 6 | 1
  Weight increased | 0 | 7 | 0
  Weight decreased | 2 | 3 | 0
  Blood pressure diastolic increased | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: from trial start on to any time before final assessment of the patient, up to 33 weeks
Arm/Group | Pramipexole Extended Release (PPX ER) | Pramipexole Immediate Release (PPX IR) | Placebo
Serious Adverse Events (participants affected / at risk) | 16/223 | 11/213 | 4/103
Other Adverse Events (participants affected / at risk) | 142/223 | 133/213 | 44/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole Extended Release (PPX ER) (N=223) | Pramipexole Immediate Release (PPX IR) (N=213) | Placebo (N=103)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Heart rate irregular (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Global amnesia (Nervous system disorders) | 0 | 1 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 1 | 0
Hallucinations, mixed (Psychiatric disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole Extended Release (PPX ER) (N=223) | Pramipexole Immediate Release (PPX IR) (N=213) | Placebo (N=103)
Constipation (Gastrointestinal disorders) | 31 | 25 | 2
Dry mouth (Gastrointestinal disorders) | 12 | 8 | 1
Nausea (Gastrointestinal disorders) | 48 | 51 | 9
Fatigue (General disorders) | 14 | 11 | 4
Oedema peripheral (General disorders) | 12 | 18 | 4
Nasopharyngitis (Infections and infestations) | 14 | 9 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 11 | 6
Dizziness (Nervous system disorders) | 26 | 25 | 7
Headache (Nervous system disorders) | 7 | 15 | 6
Somnolence (Nervous system disorders) | 81 | 70 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract